CLINICAL TRIAL: NCT02489760
Title: Etanercept Versus Adalimumab in the Treatment of Patients With Ankylosing Spondylitis. A Switch Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, GCRC, Etanercept versus Adalimumab in the Treatment of Patients with Ankylosing Spondylitis. A Switch Study., Chung Shan Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CS08019
Record Dates: First submitted 2015-06-27; First posted 2015-07-03 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Ankylosing Spondylitis
Keywords: Etanercept; Adalimumab; Ankylosing Spondylitis; Switch Study
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Adalimumab; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab switch to Etanercept (Experimental): At week 8, the treatment arm will be switched to etanercept 25 mg subcutaneously biweekly for another 8 weeks.
  Interventions: Biological: Adalimumab; Biological: Etanercept
- Etanercept switch to Adalimumab (Experimental): At week 8, the control arm will be switched to adalimumab 40 mg subcutaneously biweekly for another 8 weeks.
  Interventions: Biological: Adalimumab; Biological: Etanercept

INTERVENTIONS:
Biological: Adalimumab — The treatment arm will receive adalimumab 40 mg subcutaneously biweekly
  Other Names: Humira
Biological: Etanercept — The control arm will continue etanercept 25 mg subcutaneously twice a week
  Other Names: Enbrel

SUMMARY:
To determine the safety and efficacy of switch effects to adalimumab in etanercept-treated AS patients.

DETAILED DESCRIPTION:
This single-centre, open-labeled randomized controlled study will evaluate the safety and efficacy of adalimumab in etanercept-treated Ankylosing Spondylitis(AS) patients.

Thirty patients will be enrolled and randomized equally into two arms.

Dosage and Administration：For standard dose(etanercept 50 mg weekly) treated patients, the treatment arm will receive adalimumab 40 mg subcutaneously biweekly for 8 weeks. The control arm will continue etanercept 25 mg subcutaneously twice a week for 8 weeks. At week 8, the control arm will be switched to adalimumab 40 mg subcutaneously biweekly for another 8 weeks.For half dose(etanercept 25 mg weekly) treated patients, the treatment arm will receive adalimumab 40 mg subcutaneously monthly for 8 weeks. The control arm will continue etanercept 25 mg subcutaneously weekly for 8 weeks. At week 8, the control arm will be switched to adalimumab 40 mg subcutaneously monthly for another 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AS, as defined by 1984 Modified New York Criteria for AS.
* Stable background therapy as non-steroid anti-inflammatory for 2 weeks.
* Stable glucocorticoid for 4 weeks.
* Stable disease-modifying anti-rheumatic drugs, eg. sulphasalazine, methotrexate for 8 weeks.
* Stable anti-TNF biologics for 4 weeks.
* Written informed consent.

Exclusion Criteria:

* Serum creatinine ≥3.0 mg/dl.
* GPT≥5 times the laboratory's upper limit of normal.
* Pregnant or breast-feeding women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Bath AS disease activity index (BASDAI) | weeks 8
  The score of BASDAI on weeks 8

CONTACTS AND LOCATIONS:
Overall Officials: Wei C- C, M.D., Study Director — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Wei JC, Tsou HK, Leong PY, Chen CY, Huang JX. Head-to-Head Comparison of Etanercept vs. Adalimumab in the Treatment of Ankylosing Spondylitis: An Open-Label Randomized Controlled Crossover Clinical Trial. Front Med (Lausanne). 2020 Oct 30;7:566160. doi: 10.3389/fmed.2020.566160. eCollection 2020. PMID 33195311